CLINICAL TRIAL: NCT00684515
Title: Phase II Study of SCH 530348 in Subjects With Cerebral Infarction
Brief Title: Trial to Assess the Safety of Vorapaxar in Japanese Subjects With Cerebral Infarction (P05005; MK-5348-017)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05005
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2014-07-29 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — vorapaxar; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vorapaxar 2.5 mg + Aspirin (Experimental): Vorapaxar oral tablets; once daily for 60 days + Aspirin.
  Interventions: Drug: Vorapaxar 2.5 mg; Drug: Aspirin 75-150 mg
- Vorapaxar 1 mg + Aspirin (Experimental): Vorapaxar oral tablets; once daily for 60 days + Aspirin.
  Interventions: Drug: Vorapaxar 1 mg; Drug: Aspirin 75-150 mg
- Placebo + Aspirin (Placebo Comparator): Placebo oral tablets; once daily for 60 days + Aspirin
  Interventions: Drug: Placebo; Drug: Aspirin 75-150 mg

INTERVENTIONS:
Drug: Vorapaxar 2.5 mg — Oral tablets; once daily for 60 days.
  Arms: Vorapaxar 2.5 mg + Aspirin
Drug: Vorapaxar 1 mg — Oral tablets; once daily for 60 days
  Arms: Vorapaxar 1 mg + Aspirin
Drug: Placebo — oral tablets; once daily for 60 days
  Arms: Placebo + Aspirin
Drug: Aspirin 75-150 mg — oral tablets; once daily for 60 days

SUMMARY:
The study is designed to assess safety of Vorapaxar when added to standard of care (aspirin) in Japanese subjects with cerebral infarction. The study will assess incidence and tolerability of bleeding, major adverse cardiac events, all adverse events, and effect on expression of markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old with last cerebral infarction (excluding cardiogenic cerebral embolism) having occurred from 14 days to less than 1 year after onset (at the time of obtaining consent), with stable nervous system for more than 24 hours and known course of disease.
* Participants confirmed to have cerebral infarction lesion by brain computerized tomography (CT) or magnetic resonance imaging (MRI).
* Both of in-participant and out-participant
* Willing to give appropriate informed consent and complete all study-related procedures and able to adhere to dosing and visit schedules.
* Women of child-bearing potential (all postmenopausal women who are <1 year menopausal or who have not had surgical sterilization or a hysterectomy are considered to be women of child-bearing potential) must agree to use a medically accepted method of contraception while receiving protocol-specified study drug, and for 60 days after completion or discontinuation of the medication.

Exclusion Criteria:

* Pregnancy and nursing patients (premenopausal women should have a negative pregnancy test result confirmed before enrollment)
* Participant with any serious complication or any condition that the investigator feels that would cause a significant hazard to the participant if the study drug is administered.
* Known hypersensitivity to any component of the study drug.
* Participation in a study or use of an investigational study drug within 30 days before obtaining consent.
* Member of the staff personnel directly involved with this study
* Family member of the study staff.
* History of a bleeding diathesis, or evidence of active abnormal bleeding within 30 days before obtaining consent.
* History of cerebral hemorrhage.
* Severe hypertension (systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg).
* Major surgery within 2 weeks before obtaining consent.
* Known platelet count <100,000/mm^3
* Participants confirmed to have cerebral bleeding or any causes of cerebral bleeding by brain CT or MRI.
* Participants with transient ischemic attack (TIA), progressive stroke or cardiogenic cerebral embolism.
* Known impairment of renal function (serum creatinine >2.0 mg/dL [>176.8 (umol/L]), dysproteinemia, nephrotic syndrome, or other renal disease
* Active or chronic hepatobiliary system or hepatic disease, or aspartate aminotransferase (GOT) or alanine aminotransferate (GPT) activity more than two times greater than the upper limit of the laboratory normal range.
* Participants with contraindictation to aspirin.
* Scheduled to have PCI (peripheral coronary intervention), peripheral interventional event, carotid endarterectomy, intra- and extra- cranial bypass surgery and intravascular surgery (angioplasty) during the study period.
* Combination therapy with unfractionated heparin, tissue plasminogen activator, urokinase, warfarin, factor Xa inhibitor, direct thrombin inhibitor or antiplatelet agents other than aspirin after obtaining consent, or scheduled to have the above combination therapy.
* Any serious impairment which would make detection of new ischemic events difficult (eg, bedridden participants, participants with total nursing care, dementia participants, etc.) or consciousness disturbance which may cause aspiration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-09-21 (Actual); Primary Completion 2007-11-08 (Actual); Study Completion 2007-11-08 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Shinohara Y, Goto S, Doi M, Jensen P. Safety of the novel protease-activated receptor-1 antagonist vorapaxar in Japanese patients with a history of ischemic stroke. J Stroke Cerebrovasc Dis. 2012 May;21(4):318-24. doi: 10.1016/j.jstrokecerebrovasdis.2010.09.005. Epub 2010 Oct 14. PMID 20947374
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05005&kw=P05005&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorapaxar 1 mg: Vorapaxar 1 mg tablets administered orally once daily for 60 days.
- Vorapaxar 2.5 mg: Vorapaxar 2.5 mg tablets administered orally once daily for 60 days.
- Placebo: Matching placbo tablets to Vorapaxar administered orally once daily for 60 days.
Period: Overall Study
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Started | 33 | 29 | 28
Completed | 29 | 26 | 27
Not Completed | 4 | 3 | 1
Not completed — Adverse Event | 3 | 3 | 1
Not completed — Protocol-Defined Clinical Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo | Total
Number analyzed (Participants) | 33 | 29 | 28 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (10.0) | 65.8 (11.6) | 63.7 (8.9) | 64.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 5 | 21
  Male | 26 | 20 | 23 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Non-Major Adverse Cardiac Events (Non-MACE)
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function, or chemistry of the body temporarily associated with study drug administration, whether or not considered related to study drug. MACE events were defined as nonfatal myocardial infarction (MI), nonfatal stroke, hospitalization due to recurrent ischemia, or urgent coronary revascularization. All MACE events were excluded from this analysis.
Time Frame: Up to Day 121
Population: The population consisted of all enrolled participants that received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Number analyzed (Participants) | 33 | 29 | 28
Participants | 27 | 27 | 22

2. Secondary Outcome: Number of Paticipants Experiencing Thrombolysis in Myocardial Infarction (TIMI) Major, Minor, and Non-TIMI Bleeding Events
Description: Major TIMI bleeding was defined as any intracranial bleeding (excluding micohemorrhages <10 mm evident on magnetic resonance imaging [MRI]), clinical over signs of hemorrhge associated with a drop in hemoglobin >=5 g/dL, or fatal bleeding (bleeding that directly results in death within 7 days). Minor TIMI bleeding was defined as any clinically overt bleeding resulting in a hemoglobin drop of 3 to <5 g/dL. Non-TIMI bleeding included all bleeding events not covered under Major TIMI or Minor TIMI bleeding.
Time Frame: Up to Day 60
Population: The population consisted of all enrolled participants that received at least one dose of study drug and had TIMI bleeding data available.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Number analyzed (Participants) | 33 | 29 | 28
Participants
  Major TIMI Bleeding | 0 | 0 | 0
  Minor TIMI Bleeding | 0 | 0 | 1
  Non-TIMI Bleeding | 5 | 10 | 6

3. Secondary Outcome: Number of Participants With MACE or Death
Description: The number of participants experiencing major cardiac events or death was evaluated up to Day 121. Major cardiac events were defined as nonfatal stroke, hospitalization due to recurrent ischemia, or urgent coronary revascularization.
Time Frame: Up to Day 121
Population: The population consisted of all enrolled participants that received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Number analyzed (Participants) | 33 | 29 | 28
Participants
  MACE | 1 | 1 | 3
  Death | 0 | 0 | 0

4. Secondary Outcome: Median High-Sensitivity C-Reactive Protein (Hs-CRP) Levels By Study Visit
Description: Participant blood samples were collected to determine the median serum level of hs-CRP. hs-cRP levels reflect the underlying level of inflammation. The higher the level, the greater the disease burden.
Time Frame: Up to Day 60
Population: The population consisted of all enrolled participants who received at least one dose of study drug and had hs-CRP data available.
Measure: Median (Standard Deviation); unit: mg/L
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Number analyzed (Participants) | 33 | 29 | 28
mg/L
  Baseline (n=33, 29, 28) | 0.65 (1.44) | 0.67 (1.66) | 0.56 (1.06)
  Day 7 (n=32, 28, 27) | 0.77 (2.33) | 0.49 (0.73) | 0.41 (0.58)
  Day 14 (32, 29, 28) | 0.93 (2.69) | 0.62 (0.79) | 0.44 (0.72)
  Day 30 (n=31, 28, 28) | 0.96 (3.95) | 0.55 (1.07) | 0.56 (0.95)
  Day 45 (n=29, 27, 28) | 0.70 (1.09) | 0.48 (0.74) | 0.59 (0.76)
  Day 60 (n=29, 26, 27) | 0.59 (0.58) | 0.53 (0.63) | 0.61 (0.93)

5. Secondary Outcome: Mean CD40 Ligand Levels By Study Visit
Description: Participant blood samples were collected to determine the mean serum level of CD40 ligand. CD40 ligand values represent the level of disease activation with a higher level of CD40 ligand indicating a greater underlying risk.
Time Frame: Up to Day 60
Population: The population consisted of all enrolled participants that received at least one dose of study drug and had CD40 ligand data available.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Number analyzed (Participants) | 33 | 29 | 28
mg/L
  Baseline (n=33, 29, 28) | 6.5 (0.62) | 8.3 (0.77) | 5.9 (0.62)
  Day 7 (n=32, 28, 27) | 7.2 (0.71) | 5.8 (0.74) | 5.6 (0.60)
  Day 14 (n=32, 29, 28) | 6.3 (0.64) | 6.5 (0.79) | 6.6 (0.66)
  Day 30 (n=31, 28, 28) | 6.7 (0.79) | 7.1 (0.78) | 5.9 (0.60)
  Day 45 (n=29, 27, 28) | 5.9 (0.77) | 5.7 (0.77) | 6.2 (0.54)
  Day 60 (n=29, 26, 27) | 6.2 (0.82) | 5.3 (0.76) | 6.0 (0.56)

6. Secondary Outcome: Mean Membrane-Bound P-Selectin Levels By Study Visit
Description: Participant blood samples were collected at Baseline, Day 30, and Day 60 to determine the mean level of membrane-bound p-selectin in the serum. Membrane-bound P-selectin levels reflect the underlying level of inflammation. Intensity levels are reported in arbitrary units 0 (dark) to 1023 (bright). Higher values correspond to greater membrane-bound P-Selectin levels.
Time Frame: Up to Day 60
Population: The population consisted of all enrolled participants that received at least one dose of study drug and had membrane-bound p-selectin data available.
Measure: Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Number analyzed (Participants) | 2 | 1 | 3
Arbitrary Units
  Baseline (n=2, 1, 3) | 15.7 (0.80) | 19.5 (NA) — Due to the sample size of 1 participant, calculation of the SE was not possible. | 17.4 (1.06)
  Day 30 (n=2, 1, 3) | 19.9 (4.20) | 16.6 (NA) — Due to the sample size of 1 participant, calculation of the SE was not possible. | 17.1 (1.10)
  Day 60 (n=2, 1, 3) | 17.8 (0.05) | 18.3 (NA) — Due to the sample size of 1 participant, calculation of the SE was not possible. | 18.0 (0.07)

ADVERSE EVENTS:
Time Frame: Up to Day 121
Arm/Group | Vorapaxar 1 mg | Vorapaxar 2.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/29 | 3/28
Other Adverse Events (participants affected / at risk) | 26/33 | 24/29 | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar 1 mg (N=33) | Vorapaxar 2.5 mg (N=29) | Placebo (N=28)
Arterial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebellar Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar 1 mg (N=33) | Vorapaxar 2.5 mg (N=29) | Placebo (N=28)
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Supraventricular Extrasystoles (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Feeling Abnormal (General disorders) | 1 (1) | 2 (3) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (9) | 9 (9) | 1 (2)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 5 (5) | 2 (3) | 4 (4)
Blood Glucose Increased (Investigations) | 1 (2) | 3 (3) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood Triglycerides Increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Blood Urine Present (Investigations) | 1 (1) | 3 (3) | 2 (2)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 2 (2) | 1 (1)
Occult Blood Positive (Investigations) | 11 (12) | 10 (10) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Cerebral Infarction (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2)
Cervicobrachial Syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior approval by the Sponsor is required before the results obtained in the clinical study can be made public by the investigator (sub-investigator) in a publication or at a medical meeting.